CLINICAL TRIAL: NCT01467232
Title: Implantation of Autologous CD133+ Stem Cells in Patients Undergoing CABG
Brief Title: IMPACT-CABG Trial: IMPlantation of Autologous CD133+ sTem Cells in Patients Undergoing Coronary Artery Bypass Grafting
Acronym: IMPACT-CABG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Miltenyi Biotec, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHN-CCR-002
Record Dates: First submitted 2011-10-28; First posted 2011-11-08 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Heart Failure; Heart Attack; Coronary Artery Bypass Surgery
MeSH Terms: conditions — Heart Failure; Myocardial Infarction | interventions — AC133 Antigen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous CD133+ Stem Cells (Experimental): Autologous CD133+ stem cells
  Interventions: Biological: Injection of autologous CD133+ stem cells at the time of coronary artery bypass grafting
- Saline solution containing autologous plasma (Placebo Comparator): Saline solution containing autologous plasma without CD133+ (indistinguishable from the autologous CD133+ stem cells)
  Interventions: Biological: Injection of autologous CD133+ stem cells at the time of coronary artery bypass grafting

INTERVENTIONS:
Biological: Injection of autologous CD133+ stem cells at the time of coronary artery bypass grafting — Following completion of the distal coronary artery bypasses, autologous CD133+ stem cells, or placebo (saline solution containing autologous plasma without CD133+) will be injected into the myocardium.
  Other Names: Autologous CD133+ stem cells or placebo solution containing autologous plasma without CD133+
  Arms: Autologous CD133+ Stem Cells
Biological: Injection of autologous CD133+ stem cells at the time of coronary artery bypass grafting — Following completion of the distal coronary artery bypasses, autologous CD133+ stem cells, or placebo (saline solution containing autologous plasma without CD133+) will be injected into the myocardium
  Other Names: Autologous CD133+ stem cells or placebo solution containing autologous plasma without CD133+.
  Arms: Saline solution containing autologous plasma

SUMMARY:
Following myocardial infarct, cellular therapy is a potential approach to repopulate the injured myocardium, to treat heart failure and restore cardiac function. The purpose of this study is to assess the safety, feasibility and efficacy of intramyocardial delivery of selected autologous CD133+ bone marrow stem cells at the time of coronary artery bypass grafting in patients with chronic ischemic cardiomyopathy.

DETAILED DESCRIPTION:
CD133+ are well characterized distinct early progenitor group of stem cells that possess high engraftment, pluripotent and angiogenic capacity and proved to be valuable for cardiac repair by promoting neovascularization, inhibition of apoptosis and cardiomyogenesis.

The investigators proposed research protocol involves patients with chronic ischemic heart disease and left ventricular dysfunction undergoing coronary artery bypass grafting (CABG). In this phase II clinical trial, prospective, randomized, 2 arm, double-blind, placebo-controlled study, the investigators will assess the safety, feasibility and functional effect of intra-myocardial injection of highly selected autologous CD133+ bone marrow stem cells to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, and ≤75 years.
* Patients with severe chronic ischemic cardiomyopathy manifested by Canadian Cardiovascular Society (CCS) class II or greater angina, and/or New York Heart Association (NYHA) class II or greater dyspnea, AND who have undergone diagnostic coronary angiography demonstrating ≥70% diameter narrowing of at least two major coronary arteries or branches or ≥50% diameter narrowing of the left main coronary artery.
* Significant left ventricular systolic dysfunction evaluated by echocardiography or LV angiography (LV ejection fraction ≤45% but ≥25%) due to a prior myocardial infarction. This area of left ventricular dysfunction should be akinetic or severely hypokinetic, not dyskinetic or aneurysmal, when assessed by echocardiography or LV angiogram.
* No contraindications or exclusions (see below).
* Willingness to participate and ability to provide informed consent.

Exclusion Criteria:

* contraindications to magnetic resonance imaging (MRI) including presence of an implantable cardiac defibrillator (ICD) or permanent pacemaker (PPM), or cases in which it is anticipated that an ICD or PPM will be implanted prior to the 6 month follow-up or claustrophobia (thus precluding performance of follow-up MRI scans).
* Need for urgent or emergent revascularization.
* Anticipated for concomitant surgical procedure at the time of CABG (e.g. valve repair or replacement, aneurysm resection, etc.).
* Hemodynamically unstable patients, as defined by heart rate ≤40/min or ≥100/min, and/or systolic blood pressure <90 mmHg or ≥200 mmHg, and/or ongoing need for intravenous inotropic or vasopressor medications.
* Patients with confirmed myocardial infarction within 14 days, and/or rising cardiac biomarker proteins (i.e. CK-MB or troponin), and/or worsening ECG changes.
* Prior CABG surgery.
* Stroke within 3 months prior to plan CABG.
* Immunosuppressive medication (e.g. prednisone, cyclophosphamide, etanercept, etc.)
* Severe chronic renal insufficiency (serum creatinine ≥ 200 mmol/dl or need for dialysis),liver disease, (diagnosis of cirrhosis, chronic hepatitis, or elevated serum transaminases ≥3 times the upper limit of normal), cerebrovascular disease requiring concomitant carotid endarterectomy, peripheral arterial disease (claudication as the primary factor limiting activity), active non-dermatological malignancy requiring on-going treatment, or any other condition that would place the patient at increased risk for complications during the first 6 months after the procedure in the judgement of the attending cardiologist or cardiac surgeon.
* Contra-indication to bone marrow aspiration (Thrombocytopenia <50,000 mm3, INR >2.0 ).
* Hemoglobin less than 10g/dL, white blood cell count less than 4,000/mm3, absolute neutrophil count less than 1500/mm3
* Active infection, with a temperature greater than 37.5°C within 48 hours prior to surgery and an unexplained white blood cell count in excess of 10,000/mm3
* Myelodysplastic syndrome
* Significant cognitive impairment
* Any condition associated with a life expectancy of less than 6 months
* Known allergic reaction or contraindication to any of the components of the CD133+ enriched cells
* Participation in other studies
* History of severe ventricular tachyarrhythmia's requiring treatment
* Positive laboratory test results or a history of syphilis, Hepatitis B Virus, Hepatitis C Virus, Human T-Lymphotropic Virus Type 1 and 2, and Human Immunodeficiency Virus.
* Pregnant woman
* Inability or unwillingness to provide written informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2014-11 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Freedom from Major Adverse Cardiac Event | 6 months
  cardiac death, myocardial infarct, repeat coronary bypass grafting or percutaneous intervention of bypassed artery.
Freedom from major arrhythmia | 6 months
  sustained ventricular tachycardia or survived sudden death.

SECONDARY OUTCOMES:
Regional myocardial perfusion and function assessed by magnetic resonance scans | 6 months
Global ventricular function assessed by echocardiographic measures of ejection fraction | 6 months
Relief of symptom severity after CABG surgery | 6 months
Device performance end point | baseline
  Feasibility to produce from 100ml of bone marrow aspiration a final cell product that contains a target CD133+ cells higher than 0.5 million with a purity superior to 30% and a recovery superior to 10%.
Quality of Life after CABG surgery | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Terrence M Yau, MD, Principal Investigator — Peter Munk Cardiac Centre / University Health Network
Locations (1):
- Peter Munk Cardiac Center/ University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Noiseux N, Mansour S, Weisel R, Stevens LM, Der Sarkissian S, Tsang K, Crean AM, Larose E, Li SH, Wintersperger B, Vu MQ, Prieto I, Li RK, Roy DC, Yau TM. The IMPACT-CABG trial: A multicenter, randomized clinical trial of CD133+ stem cell therapy during coronary artery bypass grafting for ischemic cardiomyopathy. J Thorac Cardiovasc Surg. 2016 Dec;152(6):1582-1588.e2. doi: 10.1016/j.jtcvs.2016.07.067. Epub 2016 Aug 13. PMID 27665225